CLINICAL TRIAL: NCT04279444
Title: Open-Label Study to Evaluate the Effect of BKR-017 on Insulin Resistance and Other Metabolic Parameters in Type 2 Diabetes Patients
Brief Title: Effects of BKR-017 on Insulin Resistance in Type 2 Diabetes Patients
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: BioKier Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: CL-401
Record Dates: First submitted 2020-02-19; First posted 2020-02-21 (Actual); Last update posted 2020-12-04 (Actual); Status verified 2020-12

CONDITIONS: Type 2 Diabetes
MeSH Terms: conditions — Diabetes Mellitus, Type 2

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Active BKR-017 (Experimental): Open label study. All patients will receive 28 days of active treatment.
  Interventions: Dietary Supplement: BKR-017

INTERVENTIONS:
Dietary Supplement: BKR-017 — BioKier, Inc. is developing colon-targeted, oral formulations of natural gut hormone secretagogues as non-prescription medical foods or supplements for nutritional use for improvement of insulin sensitivity.

SUMMARY:
The purpose of this study is to evaluate the effect of BKR-017 on insulin resistance in type 2 diabetes (T2D) subjects during 28 days of active test product administration.

DETAILED DESCRIPTION:
The study consists of a screening period followed by a 28-day treatment period. All subjects will receive test product.

There are a total of 4 study visits including screening. Visit 1 is the screening visit. Eligible subject must have an HbA1c between 6.5 -10.5% and with HOMA-IR ≥ 2.7 (calculated from fasting insulin and fasting glucose). Visits 2 and 4 are overnight visits during which time a Mixed Meal Tolerance (MMTT) will be performed after an overnight fast. The MMTT requires an indwelling IV catheter so that 11 blood draws can be more comfortably be obtained over a period of 4 hours. At Visit 3,subjects will be evaluated and test product will be replenished. Routine chemistry and hematology testing are done and two time periods during the study and a physical exam is performed at screening

ELIGIBILITY:
Inclusion Criteria:

1. Males and females between the ages of 18 and 70 years at the time of screening, inclusive
2. Diagnosed with T2D and under the care of a healthcare professional for its management
3. HbA1c 6.5-10.5%, inclusive
4. HOMA-IR 2.7 and above
5. Has given written informed consent to participate in this study
6. Willing to complete 28-day test period, including two overnight stays
7. Willing to maintain current diet and exercise routine and current prescription medications for the duration of the study

Exclusion Criteria:

1. Type 1 diabetes
2. History of bariatric or intestinal surgery
3. Active gastrointestinal disease including but not limited to irritable bowel syndrome, inflammatory bowel disease (e.g., Crohn's disease and ulcerative colitis), diverticulitis, gastroparesis, or chronic/frequent diarrhea or chronic/frequent constipation
4. Active and clinically significant hepatic, pancreatic disease, or renal disease as determined by the investigator
5. History of significant heart disease, including congestive heart failure, prior MI, chronic atrial or ventricular fibrillation, coronary artery disease, cerebral vascular disease or other cardiovascular disease, that in the opinion of the investigator should exclude the subject from the study
6. Severely uncontrolled hypertension at screening defined as a systolic blood pressure > 180 mmHg or a diastolic blood pressure > 110 mmHg on the average of two seated measurements after being at rest for at least 5 minutes
7. Uncontrolled hyperthyroidism or hypothyroidism, or other significant thyroid disease
8. Active significant infection as determined by the investigator
9. Known allergy to butyrate or any of the components of the tablets
10. Participation in a clinical trial and/or treatment with an investigational drug during the 30 days before screening, or within 5 half-lives of receipt of an investigational drug or twice the duration of the biological effect of any investigational drug (whichever is longer)
11. Allergy or intolerance to Boost® High Protein drink
12. Pregnant, nursing, or trying to become pregnant
13. Presence of pitting edema on physical exam
14. High fiber diet
15. In the investigator's judgment, the subject is not suitable for the study for any other reason or cannot commit to the requirements of the study.
16. Subject is taking one or more of the excluded therapies. See list of excluded therapies in section 4.4.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 14 (Actual)
Dates: Start 2020-06-16 (Actual); Primary Completion 2020-11-10 (Actual); Study Completion 2020-11-15 (Actual)

PRIMARY OUTCOMES:
Insulin resistance (HOMA-IR) | 28 days of active test product administration
  Changes, Day 0 to Day 28 in patient's insulin resistance (HOMA-IR)

SECONDARY OUTCOMES:
Fasting glucose | Day 0 to Day 28
  Changes in fasting glucose
Fasting insulin | Day 0 to Day 28
  Changes in fasting insulin
Fasting triglycerides | Day 0 to Day 28
  Changes in fasting triglycerides
Triglyceride, glucose, and insulin AUCs | 4 hours in the MMTT
  Changes in triglyceride, glucose, and insulin AUCs

CONTACTS AND LOCATIONS:
Overall Officials: George Szewczyk, PhD, Study Chair — BioKier Inc.
Locations (1):
- Pennington Biomedical Research Center, Baton Rouge, Louisiana, United States

IPD SHARING:
Plan to Share IPD: No